CLINICAL TRIAL: NCT04274725
Title: Managing the Experience of Prostate Biopsy: What Are Men's Perceptions of Their Lived Experience and Support Needs
Brief Title: Men's Experience of Prostate Biopsy
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR: 4964
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Prostate Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Men aged over 18 having a first or second diagnostic prostate biopsy at the Royal Marsden NHS Foundation Trust or Epsom General Hospital may be invited to take part in one to one interview within 6 months of having the procedure done to talk about their experience

DETAILED DESCRIPTION:
Men aged over 18 having a first or second diagnostic prostate biopsy at the Royal Marsden NHS Foundation Trust or Epsom General Hospital will be approached by their Urology team or study Researcher with an information sheet about the study pre or post biopsy. The participant information sheet outlines that the study will involve being interviewed by the researcher, Kathryn Myhill as part of her doctoral research and being asked about their perceptions of their biopsy experience and what it was like to go through it. Men who return an expression of interest reply slip by post will be contacted by the researcher or they can contact her directly via the email or phone details given in the PIS. The researcher will answer any queries about the study and explore whether they would like to take part in an interview. A one to one interview will then be offered in a non-clinical, private room at the hospital where their biopsy took place (Royal Marsden Hospital, Epsom General Hospital) or at their workplace or home.

ELIGIBILITY:
* Inclusion Criteria:
* Men aged over 18 having a first or second diagnostic prostate biopsy at either the Royal Marsden NHS Foundation Trust or Epsom General Hospital
* Within 6 months of their prostate biopsy being done
* Exclusion Criteria:
* Men unable to give informed consent/ men needing a translator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Men aged over 18
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
To review the experience of prostate biopsy | two years
  Qualitative evaluation of biopsy experience

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Epsom General Hospital, London
  - Royal Marsden NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No